CLINICAL TRIAL: NCT03732794
Title: AtriCure CryoICE Lesions for Persistent and Long-standing Persistent Atrial Fibrillation Treatment During Concomitant On-Pump Endo/Epicardial Cardiac Surgery
Brief Title: AtriCure CryoICE Lesions for Persistent and Long-standing Persistent Atrial Fibrillation Treatment
Acronym: ICE-AFIB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2018-1
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation (AF); Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AtriCure CryoICE & AtriClip LAA Exclusion (Experimental): AtriCure CryoICE system performing the Cox-Maze III lesion set, in conjunction with LAA exclusion using the AtriClip device.
  Interventions: Device: AtriCure CryoICE & AtriClip LAA Exclusion

INTERVENTIONS:
Device: AtriCure CryoICE & AtriClip LAA Exclusion — AtriCure CryoICE system in performing the Cox-Maze III lesion set, in conjunction with LAA exclusion using the AtriClip device.

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of the AtriCure CryoICE system in performing the Cox-Maze III lesion set, in conjunction with Left Atrial Appendage (LAA) exclusion using the AtriClip device.

DETAILED DESCRIPTION:
The AtriCure CryoICE Ablation System is being studied to ablate cardiac tissue during surgery for the treatment of Persistent and Long-standing Persistent atrial fibrillation in open concomitant cardiac surgery.

The effectiveness of the device will be demonstrated by establishing that the device effectively eliminates persistent and long-standing persistent atrial fibrillation in a clinically significant proportion of treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age
2. Subject has history of persistent or long-standing persistent atrial fibrillation as defined by the 2017 Heart Rhythm Society (HRS)/European Heart Rhythm Association (EHRA)/ European Cardiac Arrhythmia Society (ECAS) Guidelines
3. Stable Subject that is scheduled to undergo non-emergent cardiac surgical procedure(s) to be performed on cardiopulmonary bypass including open-heart surgery for one or more of the following: Mitral valve repair or replacement, Aortic valve repair or replacement, Tricuspid valve repair or replacement, and Coronary artery bypass procedures
4. Left Ventricular Ejection Fraction ≥ 30% (determined by echocardiography or cardiac catheterization performed within 60 days of enrollment as documented in patient medical history)
5. Subject is willing and able to provide written informed consent
6. Subject has a life expectancy of at least 5 years
7. Subject is willing and able to return for scheduled follow-up visits.

Exclusion Criteria:

1. Stand-alone AF without indication(s) for concomitant Coronary Artery Bypass Graft (CABG) and/or valve surgery
2. Previous surgical Maze procedure
3. Wolff-Parkinson-White syndrome or other Supra-Ventricular arrhythmia, Atrioventricular (AV) nodal reentry
4. Prior cardiac surgery (Redo)
5. Subjects requiring surgery other than CABG and/or cardiac valve surgery and/or patent foramen ovale repair, and/or atrial septal defect repair.
6. Class IV New York Heart Association (NYHA) heart failure symptoms
7. Prior history of cerebrovascular accident within 6 months or at any time if there is residual neurological deficit
8. Documented ST-segment elevation Myocardial Infarction (MI) within the 6 weeks prior to study enrollment
9. Need for emergent cardiac surgery (i.e. cardiogenic shock)
10. Known carotid artery stenosis greater than 80%
11. Documented AF duration of greater than ten years
12. LA diameter >7 cm by Transthoracic echocardiography (TTE)
13. Current diagnosis of active systemic infection
14. Severe peripheral arterial occlusive disease defined as claudication with minimal exertion
15. Renal failure requiring dialysis or hepatic failure
16. A known drug and/or alcohol addiction
17. Mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study
18. Pregnancy or desire to get pregnant within 12-months of the study treatment
19. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
20. Requires anti-arrhythmic drug therapy for the treatment of a ventricular arrhythmia
21. Subjects who have been treated with thoracic radiation
22. Subjects in current chemotherapy
23. Subjects on long term treatment with oral or injected steroids (not including intermittent use of inhaled steroids for respiratory diseases)
24. Subjects with known connective tissue disorders
25. Subjects with known hypertrophic obstructive cardiomyopathy
26. Subjects with known cold agglutinin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Freedom from AF/Atrial Flutter (AFL)/Atrial Tachycardia (AT) | 12 months
  Freedom from AF/AFL/AT lasting >30 seconds in duration 6 through 12-months following the ablation procedure in the absence of Class I or III antiarrhythmic drugs (AADs).
Safety Endpoint: composite acute major adverse event (MAE) rate | 30 days
  The composite acute major adverse event (MAE) rate, within 30-days post-procedure and deaths after 30-days if death is procedure related.

SECONDARY OUTCOMES:
Composite post-procedure MAE rate (Safety). | 12 months
  Long-term safety based on MAE rate at 12-months post-procedure
Pacemaker implantation (Safety). | 12 months
  Percentage of implantation of a permanent pacemaker either in the operative period (<30 days postoperative) or at any time during follow-up period.
Overall Serious Adverse Event (SAE) rate (Safety) | 12 months
  Long-term safety based on SAE rate at 12-months post-procedure
Freedom from AF/AFL/AT in presence of previously failed Class I or III AADs (Effectiveness) | 12 months
  Freedom from AF/AFL/AT lasting >30 seconds in duration 12-months following the ablation procedure in presence of previously failed Class I or III AADs.
Freedom from AF/AFL/AT regardless of Class I or III AADs (Effectiveness) | 12 months
  Freedom from AF/AFL/AT lasting >30 seconds in duration 12-months following the ablation procedure regardless of Class I or III AADs.
Atrial Fibrillation Effect on Quality-of-Life (AFEQT) Score (Effectiveness) | 12 months
  Based on composite score (0-100). A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
  AFEQT Evaluates Health Related Quality of Life (HRQoL) across three domains Symptoms - Four questions specifically targeted to assess AF related symptoms Daily Activities - Eight questions that evaluate daily function in AF patients Treatment Concerns - Six questions that assess AF treatment concerns in patients The overall composite score and domains will be summarized by presenting the means, medians, standard deviations, interquartile ranges, minimum, and maximum
Acute procedural success (Effectiveness) | Intra-operative period
  Absence of AF at end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Washington Adventist Hospital
Locations (15):
- United States (15):
  - UCLA Medical Center, Los Angeles, California
  - Washington Adventist Hospital, Washington D.C., District of Columbia
  - Northwestern Medicine, Chicago, Illinois
  - Franciscan Health, Indianapolis, Indiana
  - Deaconess Gateway Hospital, Newburgh, Indiana
  - University Of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Mount Sinai Icahn School of Medicine, New York, New York
  - NYP-Weill Cornell, New York, New York
  - Northwell Health Systems, New York, New York
  - St. Joseph Hospital Health Center, Syracuse, New York
  - St Thomas West Hospital, Nashville, Tennessee
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, Statistical Analysis Plan (SAP), and Informed Consent (ICF) will be shared at the completion of the study.
Time Frame: Information will be available in accordance with clinical trials.gov requirements.
Access Criteria: Publicly available through clinical trials.gov